CLINICAL TRIAL: NCT01380249
Title: Phase I Study, Open, Dose Escalation, in Adult Patients With Advanced Solid Tumours, to Evaluate Tolerability, Pharmacokinetics and Pharmacodynamics of PDM08 Administered Twice a Week Cycles of 4 Weeks.
Brief Title: PDM08 Clinical Trial in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prodimed S.A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-017133-21
Record Dates: First submitted 2011-05-31; First posted 2011-06-27 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Malignant Solid Tumours
Keywords: Phase I; Phase I multiple doses; PDM08; Cancer Treatment; Pharmacokinetics and Pharmacodynamics; Advanced Solid Tumors; Prodimed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PDM08 (Experimental): To assess the tolerability and safety of increasing multiple doses administration of PDM08: 560 μg, 1.12 mg, 2.24 mg, 3.5 mg and 14 mg, 28 mg and 56 mg administered twice a week for four weeks in patients with advanced solid tumours for which there is no standard therapy or the patient is refractory to it.
  Interventions: Drug: PDM08

INTERVENTIONS:
Drug: PDM08 — To assess the tolerability and safety of increasing multiple doses administration of PDM08: 560 μg, 1.12, 2.24, 3.5, 14, 28 and 56 mg administered twice a week for four weeks in patients with advanced solid tumours for which there is no standard therapy or they are refractory to it.
  Other Names: 4-amino-5-oxo-4(pyridinium-1-ylmethyl)proline D-cis; 3S,5R-1-(3-Amino-5-carboxy-2-oxopyrrolidin-3-ylmethyl)pyridinium bromide hidrobromide

SUMMARY:
This phase I study in adult patients with advanced solid tumours is designed to evaluate toxicity, drug exposure (pharmacokinetics) and drug action (pharmacodynamics) of a new molecule, PDM08, administered twice a week cycles of 4 weeks. This drug has shown antitumoral activity in several murine cancer models.

DETAILED DESCRIPTION:
Phase I study, open, dose escalation, in adult patients with advanced solid tumours, to evaluate tolerability, pharmacokinetics and pharmacodynamics of ascending PDM08 doses administered twice a week cycles of 4 weeks.

After checking the safety of the first drug doses, a new dose escalation was proposed and approved by the Ethic Committee and the Medicines Agency.

This clinical trial is carried out in adult patients with advanced solid tumours whose disease has progressed despite standard therapy, or for which there is no standard antineoplastic therapy, or are refractory to it.

In pharmacodynamic non clinical studies, PDM08 presented antitumour activity against different tumour models including, renal, colon, lung, prostate and breast cancer models.

ELIGIBILITY:
Inclusion Criteria:

* Population: Adult patients with advanced solid tumours whose disease has progressed despite standard therapy, or for which there is no standard antineoplastic therapy, or are refractory to it.
* Informed consent must be obtained for each patient, in accordance with the guideline for Good Clinical Practice (GCP) of the International Conference of Harmonization (ICH) and with the local requirements.
* Malignant tumour, histologically or cytologically demonstrated.
* Patients age equal or greater than 18 years.
* Patients must not have an ECOG>2 (ECOG 2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours)
* The life expectancy of the patient should be superior to 3 months.
* Bilirubin<1,5 times the laboratory upper limit.
* AST and ALT less than 2,5 times the laboratory upper limit, In case of liver metastases to a value less than 5 times the laboratory upper limit.
* Women in fertile age: a pregnant test must be carried out.
* Men and women in fertile age must commit to to practice one method of birth control during their participation in the trial, and 30 days after the administration of the last dose of the experimental drug.
* The patient should have renal function parameters (creatinine) not exceeding 1.5 times the normal upper limit.
* The patient must present a hemoglobin > 9 mg/dL.
* The patient must show basal platelet count > 100.000 /mm3.
* Specific criteria:
* Patients included in the expansion cohort must present a measurable disease by RECIST criteria 1.1, and disease progression in the last 6 months.
* Patients who agree to enter into the pharmacodynamic tumour tissue substudy should present accessible tissue to carry out the biopsy safely.

Exclusion Criteria:

* Patients who have received chemotherapy, radiotherapy, immunotherapy or investigational drugs for their disease within 4 weeks prior to PDM08 first dose.
* Patients who have had surgery within 4 weeks before treatment.
* Patients with untreated brain metastases.
* Patients who are pregnant or breast-feeding.
* Those patients who present an intercurrent non-controlled disease including, but not limited to, active infections, cicatrization problems, congestive heart failure, unstable angina, cardiac arrhythmia, pulmonary disease with non controlled symptoms, non controlled psychiatric disorders or social situations that may affect the compliance with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number and grade of adverse events by participant related to PDM08. | 6 weeks for each cohort.
  Drug safety will be measured by the number and grade of adverse events, by participant, related to the drug in study (PDM08) in the cohorts studied: 560 μg, 1.12 mg, 2.24 mg, 3.5 mg and 14 mg, 28 mg and 56 mg administered twice a week for four weeks.
  The drug will be administered twice a week for four weeks.
  Safety and tolerability will be measured considering the adverse events occurred, by participant, related with the drug in study, PDM08, at each cohort.
Dose limiting toxicity (DLT) | 6 weeks.
  Drug tolerability will be assessed by determining the DLT. It will be determined for each cohort (increasing multiple doses of PDM08): 560 μg, 1.12 mg, 2.24 mg, 3.5 mg and 14 mg, 28 mg and 56 mg administered twice a week for four weeks). Dose Limiting Toxicity will be considered the dose that produces adverse events of a severity grade 3 or greater, related to the drug in study (PDM08) in the classification specified in the list of Toxicity Criteria of the National Cancer Institute (CTCAE v04.03).

SECONDARY OUTCOMES:
AUC | 4 weeks
  Blood sampling collected on Day 1 and 25 of each cohort cycle.Cohorts (doses): 560 μg, 1.12 mg, 2.24 mg, 3.5 mg and 14 mg, 28 mg and 56 mg administered twice a week for four weeks.
  Blood collection scheme: - Dose of 560 μg and 1.12 mg: 0,0.25, 1, 2, 4, 8, 12 hours post-dose, on day 1 and day 25 of each cycle. - Doses of 2.24 mg, 3.5 mg, 14 mg, 28 mg, and 56 mg: 0,0.25, 1, 2, 4, 8, 12, 16 and 24 hours post-dose, on day 1 and day 25 of each cycle.
  Pharmacokinetic parameters will be expressed as mean ± standard deviation and confidence interval 95%. Linearity will be analyzed.
Cmax | 4 weeks
  Blood sampling will be collected on Day 1 and Day 25 of each cohort cycle.Cohorts(doses): 560 μg, 1.12 mg, 2.24 mg, 3.5 mg and 14 mg, 28 mg and 56 mg administered twice a week for four weeks.
  Blood collection scheme:
  * Dose of 560 μg and 1.12 mg: 0,0.25, 1, 2, 4, 8, 12 hours post-dose, on day 1 and day 25 of each cycle.
  * Dose of 3.5 mg and 14 mg, 28 mg and 56 mg: 0,0.25, 1, 2, 4, 8, 12, 16 and 24 hours post-dose, on day 1 and day 25 of each cycle.
  Pharmacokinetic parameters will be expressed as mean ± standard deviation and confidence interval 95%. Linearity will be analyzed.
Volume of distribution (Vd) | 4 weeks
  Blood sampling will be collected on Day 1 and Day 25 of each cohort cycle.Cohorts(dose): 560 μg, 1.12 mg, 2.24 mg, 3.5 mg and 14 mg, 28 mg and 56 mg administered twice a week for four weeks.
  Blood collection scheme:
  * Dose of 1.12 mg and 2.24 mg: 0,0.25, 1, 2, 4, 8, 12 hours post-dose, on day 1 and day 25 of each cycle.
  * Dose of 2.24 mg; 3.5 mg and 14 mg, 28 mg and 56 mg: 0,0.25, 1, 2, 4, 8, 12, 16 and 24 hours post-dose, on day 1 and day 25 of each cycle.
  Pharmacokinetic parameters will be expressed as mean ± standard deviation and confidence interval 95%. Linearity will be analyzed.
Plasma half-life of PDM08 (T ½) | 4 weeks
  Blood sampling will be collected on Day 1 and Day 25 of each cohort cycle.Cohorts(dose): 560 μg, 1.12 mg, 2.24 mg, 3.5 mg and 14 mg, 28 mg and 56 mg administered twice a week for four weeks.
  Blood collection scheme:
  * Dose of 560 μg and 1.12 mg: 0,0.25, 1, 2, 4, 8, 12 hours post-dose, on day 1 and day 25 of each cycle.
  * Dose of 2.24 mg, 3.5 mg and 14 mg, 28 mg and 56 mg: 0,0.25, 1, 2, 4, 8, 12, 16 and 24 hours post-dose, on day 1 and day 25 of each cycle.
  Pharmacokinetic parameters will be expressed as mean ± standard deviation and confidence interval 95%. Linearity will be analyzed.
Changes in tumour size by Computed Tomography (CT) | 6 weeks
  Changes in tumour size will be measured by CT (RECIST criteria v.1.1) at each cohort on days 1, 4, 11, 25, 29 and 43 of the study.
  Pharmacodynamic parameters will be tabulated as raw values and sorted by dose. Statistical analysis will be performed using ANOVA with repeated measures, including baseline values as cofactor.
Tumour activity: Positron emission tomography (PET) | 6 weeks
  Changes in tumour activity will be measured by PET in each cohort on days 1, 4 11, 25, 29 and 43 of the study.
  Pharmacodynamic parameters will be tabulated as raw values and sorted by dose. Statistical analysis will be performed using ANOVA with repeated measures, including baseline values as cofactor.
Myeloid cells in peripheral blood. | 6 weeks
  Myeloid cells in peripheral blood (total myeloid cells, monocyte-macrophage series, granulocytes and myeloid suppressor in peripheral blood) will be measured in each cohort on days 1, 4, 11, 25, 29 and 43 of the study.
B and T lymphocytes and NK cells Populations | 6 weeks
  In order to determine the function of these populations the exresion of membrane markers will be analyze; and membrane markers displayed in relation to the degree of activation of lymphocytes. These parameters will be measured at each cohort on days 1, 4, 11, 25, 29 and 43 of the study.
Serum Immunoglobulins | 6 weeks
  Serum Immunoglobulins and subtypes (IgG1, IgG2, IgG3, IgG4, IgM, IgA) will be measured at each cohort on days 1, 4, 11, 25, 29 and 43 of the study.
Complement components: C3 and C4; and C-Reactive Protein (CRP) | 6 weeks
  C3 and C4 components of the complement system, CRP, and the total activity of the classical complement pathway. measured as haemolytic capacity CH50,will be measured in serum of all the participants at each cohort on days 1, 4, 11, 25, 29 and 43 of the study.
Serum cytokines | 6 weeks
  Serum cytokines that will be measured will be:IL1α, IL1β, IL2, IL4, IL5, IL6, IL7, IL10, IL12, IL17, TNFα, IFNγ, G-CSF, GM-CSF, VEGF. Serum cytokines will be measured in serum at each cohort on days 1, 4, 11, 25, 29 and 43 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Barriuso, MD, PhD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain